CLINICAL TRIAL: NCT01372007
Title: Influence of Somatuline Autogel 120mg on Post-operative Drainage After Total Mesorectum Excision for Rectumcarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/267
Record Dates: First submitted 2011-06-08; First posted 2011-06-13 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Rectal Carcinoma
Keywords: Rectal carcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lanreotide Autogel 120mg (Experimental)
  Interventions: Drug: Lanreotide Autogel 120mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanreotide Autogel 120mg — Drain fluid will be checked for hematocrit daily post-surgery. Once hematocrit levels of the drain fluid are <10%, study medication (0.246mg lanreotide base/mg solution) will be administered. After administration the volume of the drain fluid will be measured every 12 hours for at least 5 days. A sample of the drain fluid will be collected every 24 hours for at least 5 days and frozen at -70°C for total protein content, sodium and chloride analysis afterwards.
  Arms: Lanreotide Autogel 120mg
Drug: Placebo — Drain fluid will be checked for hematocrit daily post-surgery. Once hematocrit levels of the drain fluid are <10%, placebo (Sodiumchloride 0,9% 1 ampoule) will be administered. After administration the volume of the drain fluid will be measured every 12 hours for at least 5 days. A sample of the drain fluid will be collected every 24 hours for at least 5 days and frozen at -70°C for total protein content, sodium and chloride analysis afterwards.
  Arms: Placebo

SUMMARY:
Total mesorectal excision (TME) is a precise dissection of the rectum and all para-rectal lymph nodes within the mesorectal envelope. It is becoming universally recognized and accepted as the standard technique for surgical excision of rectum carcinomas. TME results in lowest rates of local recurrence, especially when combined with pre-operative chemo-radiotherapy.

Especially after pre-operative chemo-radiotherapy, the post-operative drainage may be important. The quick decrease of this drainage will enable the early mobilisation of the patient and may shorten the time of hospitalization. If this decrease in fluid production can be achieved, it will have a positive effect on the Quality of Life of the patient and will ensure health economic savings by reduction of hospitalization time and resources.

Somatostatin analogues have shown to be able to decrease the secretion of numerous types of bodily fluids.

The aim of this study is to investigate if lanreotide Autogel 120mg is capable to reduce the fluid discharge in patients that underwent a TME for rectumcarcinoma.

Lanreotide Autogel 120mg compared to placebo, administered post-surgery on the fluid discharge in the drain of the patient that underwent a total mesorectum excision (TME) for rectal carcinoma. Patient planned to have a TME will be asked to participate in the study. When they have provided written informed consent, they will be randomized 1:1 to receive either placebo or lanreotide autogel 120mg. Drain fluid will be checked for hematocrit daily post-surgery. Once hematocrit levels of the drain fluid are <10%, study medication or placebo will be administered. After administration the volume of the drain fluid will be measured every 12 hours for at least 5 days. A sample of the drain fluid will be collected every 24 hours for at least 5 days and frozen at -70°C for total protein content, sodium and chloride analysis afterwards. If the patient has a hematocrit >10% in his drain fluid for a period of 5 days, this patient can not be randomized.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients
* 18-75 years
* written informed consent to participate the study
* scheduled to have a total mesorectal excision (TME) for rectumcarcinoma

Exclusion Criteria:

* patients with a known intolerance for somatostatin analogues, lanreotide or any of it's excipients
* patients younger than 18 years
* patients unable to provide written informed consent
* patients who received somatostatin or any of it's analogues the last 30 days before the start of the study
* Pregnant and breast-feeding women
* Women not using contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
% reduction in drain fluid volume over a period of 5 days post study treatment administration in both arms. | Drain fluid will be checked every day with a minimum of 5 days or until the drain is removed.
  Drain fluid will be checked for hematocrit daily post-surgery. Once hematocrit levels of the drain fluid are <10%, study medication or placebo will be administered. After administration the volume of the drain fluid will be measured every 12 hours for at least 5 days. A sample of the drain fluid will be collected every 24 hours for at least 5 days and frozen at -70°C for total protein content, sodium and chloride analysis afterwards.

SECONDARY OUTCOMES:
Evaluation of the Quality of life of the patient. | This will be evaluated during a hospitalization of approximately 10 days.
  Patient observation to evaluate Quality of life of the patient, and time of mobilisation after surgery. Evaluation of the results and the effect on the Health economy.
Evaluation of the time of mobilisation after surgery. | This will be evaluated during a hospitalization of approximately 10 days.
  Patient observation to evaluate time of mobilisation after surgery. Evaluation of the results and the effect on the Health economy.

CONTACTS AND LOCATIONS:
Overall Officials: Piet Pattyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Universital Hospital Ghent, Ghent, Belgium